CLINICAL TRIAL: NCT02472171
Title: Suppression of Postprandial Monocyte Activation by Fruit Rich in Anti-inflammatory Polyphenols or Docosahexaenoic Acid in Humans
Brief Title: Suppression of Postprandial Monocyte Activation by Blueberries or Docosahexaenoic Acid in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 537073; 2013-03477 (Other Grant/Funding Number: National Institute of Food and Agriculture)
Record Dates: First submitted 2015-06-04; First posted 2015-06-15 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Inflammation
Keywords: n-3 polyunsaturated fatty acids; blueberries
MeSH Terms: conditions — Inflammation | interventions — Sunflower Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Experimental): Order of treatments:
  A. High saturated fat meal, placebo powder and sunflower oil B. High saturated fat meal, blueberry powder and sunflower oil C. High saturated fat meal, placebo powder and DHA
  Interventions: Dietary Supplement: High saturated fat meal, placebo powder and sunflower oil; Dietary Supplement: High saturated fat meal, blueberry powder and sunflower oil; Dietary Supplement: High saturated fat meal, placebo powder and DHA
- Group 2 (Experimental): Order of treatments:
  A. High saturated fat meal, placebo powder and sunflower oil C. High saturated fat meal, placebo powder and DHA B. High saturated fat meal, blueberry powder and sunflower oil
  Interventions: Dietary Supplement: High saturated fat meal, placebo powder and sunflower oil; Dietary Supplement: High saturated fat meal, blueberry powder and sunflower oil; Dietary Supplement: High saturated fat meal, placebo powder and DHA
- Group 3 (Experimental): Order of treatments:
  B. High saturated fat meal, blueberry powder and sunflower oil A. High saturated fat meal, placebo powder and sunflower oil C. High saturated fat meal, placebo powder and DHA
  Interventions: Dietary Supplement: High saturated fat meal, placebo powder and sunflower oil; Dietary Supplement: High saturated fat meal, blueberry powder and sunflower oil; Dietary Supplement: High saturated fat meal, placebo powder and DHA
- Group 4 (Experimental): Order of treatments:
  B. High saturated fat meal, blueberry powder and sunflower oil C. High saturated fat meal, placebo powder and DHA A. High saturated fat meal, placebo powder and sunflower oil
  Interventions: Dietary Supplement: High saturated fat meal, placebo powder and sunflower oil; Dietary Supplement: High saturated fat meal, blueberry powder and sunflower oil; Dietary Supplement: High saturated fat meal, placebo powder and DHA
- Group 5 (Experimental): Order of treatments:
  C. High saturated fat meal, placebo powder and DHA B. High saturated fat meal, blueberry powder and sunflower oil A. High saturated fat meal, placebo powder and sunflower oil
  Interventions: Dietary Supplement: High saturated fat meal, placebo powder and sunflower oil; Dietary Supplement: High saturated fat meal, blueberry powder and sunflower oil; Dietary Supplement: High saturated fat meal, placebo powder and DHA
- Group 6 (Experimental): Order of treatments:
  C. High saturated fat meal, placebo powder and DHA A. High saturated fat meal, placebo powder and sunflower oil B. High saturated fat meal, blueberry powder and sunflower oil
  Interventions: Dietary Supplement: High saturated fat meal, placebo powder and sunflower oil; Dietary Supplement: High saturated fat meal, blueberry powder and sunflower oil; Dietary Supplement: High saturated fat meal, placebo powder and DHA

INTERVENTIONS:
Dietary Supplement: High saturated fat meal, placebo powder and sunflower oil — High saturated fat meal with a blueberry flavored shake and sunflower oil
Dietary Supplement: High saturated fat meal, blueberry powder and sunflower oil — High saturated fat meal with blueberry powder shake and sunflower oil
Dietary Supplement: High saturated fat meal, placebo powder and DHA — High saturated fat meal with a blueberry flavored shake and DHA

SUMMARY:
The overall goal of the research study is to determine whether a high-fat meal causes postprandial (after meal) inflammation, and whether eating n-3 polyunsaturated fatty acids (PUFAs) or blueberries that are rich in anti-inflammatory polyphenols suppress the inflammation in healthy people.

DETAILED DESCRIPTION:
Chronic inflammation is one of the key etiological conditions associated with the development and progression of chronic diseases including Alzheimer's disease, atherosclerotic cardiovascular disease, insulin resistance, obesity and cancer. The causes of chronic inflammation and the role of diet in suppressing inflammation are challenging research questions. Pattern recognition receptors (PRRs), including Toll-like receptors (TLRs), nucleotide-binding oligomerization domain proteins (NODs), and the inflammasome expressed in innate immune cells can be activated by a variety of endogenous molecules derived from tissue injury and diet (in particular saturated fatty acids), eliciting inflammation. Dysregulated induction of PRR-mediated inflammation is known to promote the development of chronic diseases. Previous studies showed that saturated fatty acids can activate toll-like receptor 4 (TLR4) and nucleotide-binding oligomerization domain 2 (NOD2) mediated signaling pathways, whereas, docosahexaenoic acid (DHA), an n-3 polyunsaturated fatty acid, and certain polyphenols (quercetin, luteolin, Epigallocatechin gallate (EGCG), resveratrol) rich in certain fruits and vegetables inhibit TLR4 or NOD2-mediated inflammation. In addition, numerous studies have demonstrated that TLR4 knockout mice were protected from high saturated fat diet-induced inflammation and insulin resistance, suggesting that high fat diet-induced inflammation and insulin resistance are at least partly mediated through the activation of TLR4. Direct evidence of saturated fatty acids derived from a high fat meal activating PRRs in humans has not been demonstrated. Thus, the investigators propose to determine whether saturated fatty acids derived from a high saturated fat meal activate blood monocytes through PRRs and whether dietary DHA and freeze-dried blueberry powder can suppress high saturated fat meal-induced inflammation by inhibiting PRR activation.

The experimental procedures and the study activities will last for approximately 9 weeks. There will be three test days, scheduled 4 weeks apart. On the test days there will be four blood draws (one fasting blood draw and three postprandial blood draws at 1-hour, 3-hour and 6-hour after breakfast, respectively). Three endothelial function measurements (EndoPAT) will be carried out each test day. A pre-test dinner meal will be provided to the subject to eat the night before each test day. Subjects will be asked to follow and record a low antioxidant and polyphenol diet of their own choosing for 3 days prior to each test day. This includes minimizing tea, wine, coffee, chocolate, fruits, vegetables, whole grains, soy, herbs, spices, condiments, and fatty fish. All volunteers will participate in all test days, receiving in randomize cross-over fashion the following treatments:

A. High saturated fat diet, placebo powder, sunflower oil. B. High saturated fat diet, blueberry powder, sunflower oil. C. High saturated fat diet, placebo powder, DHA.

The high saturated fat meal will be identical in all treatments and may contain tortilla, cheddar cheese, beef sausage, scrambled eggs, and a smoothie style drink containing sugar, vanilla extract, oil, whole milk yogurt and the ingredients for masking treatments. The placebo powder may contain Beneprotein® (Nestlé Nutrition), Benefiber® (Novartis), oil, sugar, artificial food-grade blueberry flavor, and artificial food-grade blue and red colors. The blueberry powder (equivalent to four 1/2 cup servings) will be obtained from the U.S. Highbush Blueberry Council (Folsom, CA). The DHA will be obtained from Martek Biosciences. Blueberry or placebo powder and the DHA or sunflower oil will be combined into a blueberry flavored smoothie style drink. Neither the study subjects or the investigators will know which treatment is provided on which test day.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index of 18-25 kg/m2
* Complete Blood Count (CBC) within normal limits
* Blood chemistry panel within normal limits

Exclusion Criteria:

* following a vegetarian diet
* smoke or use tobacco products
* consume more than one alcoholic beverage per day (defined as 1 oz. distilled liquor, 3 oz. wine, or 12 oz. beer)
* taking any cholesterol lowering
* taking blood pressure medication
* taking non-steroidal anti-inflammatory drugs (NSAIDS) more than once a week and for 3 days before each test day
* taking steroids for asthma or other inflammatory states
* taking thyroid-regulating drugs
* taking over-the-counter weight loss products
* allergies or sensitivities to foods or ingredients in the test meals, especially blueberries or DHA
* taking fish or algae oil or other dietary supplements and unwilling to stop the supplements for the duration of the study (multivitamin is OK)
* Women who are pregnant, lactating or planning a pregnancy
* fasting blood cholesterol greater than 240 mg/dL
* fasting blood triglyceride greater than 300mg/dL
* hemoglobin less than 11.5 mg/dL
* blood pressure greater than 140/90 mmHg
* metabolic diseases such as diabetes mellitus, hypothyroidism, kidney disease, liver disease, bleeding disorders, autoimmune diseases, other inflammatory disease, or cancer unless greater than 5 years remission

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2015-06; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in Monocyte activation in whole blood | Measured at 0, 1, 3, and 6 hours after high fat meal with blueberries, DHA or placebo
  Change in monocyte activation using monocyte activation assay in whole blood.

SECONDARY OUTCOMES:
Change in surface markers for monocyte activation | Measured at 0, 1, 3, and 6 hours after high fat meal with blueberries, DHA or placebo
  Surface markers for monocyte activation will be measured by flow cytometry. Surface markers may include cluster of differentiation (CD) 14 (CD14), CD11c, CD11b and CD62 Ligand (CD62L) to assess monocyte activation and M1 and M2 macrophage marker proteins.
Change in systemic inflammation | Measured at 0, 1, 3, and 6 hours after high fat meal with blueberries, DHA or placebo
  Inflammatory mediators measured in whole blood or blood plasma. Inflammatory mediators include cytokines such as Interleukin-1β, Tumor Necrosis Factor-alpha, Interferon-gamma, Interleukin-6, Interleukin-8, Th1, Th2 and Th17.
Change in systemic inflammation measured indirectly | Measured at 0, 3, and 6 hours after high fat meal with blueberries, DHA or placebo
  The magnitude of the inhibition of cytokine production after 24 hour incubation of whole blood by endotoxin inhibitor, polymyxin B (PMB), is measured as an indirect assessment of endotoxin concentration. Cytokine concentrations in whole blood after 24 hour incubation with lipoprotein lipase and PMB is used to assess whether increased concentrations of non-esterified fatty acids (NEFA) and saturated fatty acids stimulate cytokine production.
Change in gene expression profile in whole blood | Measured at 0, 1, 3, and 6 hours after high fat meal with blueberries, DHA or placebo
  Gene expression measured using RNA sequencing
Change in blood lipids | Measured at 0, 1, 3, and 6 hours after high fat meal with blueberries, DHA or placebo
  Lipids, total non-esterified fatty acids, and individual fatty acids measured in blood
Change in endothelial function measurements | Measured at 0, 3, and 6 hours after high fat meal with blueberries, DHA or placebo
  Endothelial function measurements will be made using the EndoPAT system, a noninvasive endothelial function assessment tool based on peripheral arterial tone (PAT) signal technology. The change in arterial tone is elicited by creating a hyperemic response induced by local ischemia (by occlusion of the brachial artery for five minutes). The endothelial function is expressed as a Reactive Hyperemia Index as described in the manufacturer's manual.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Hwang, PhD, Principal Investigator — USDA, ARS, Western Human Nutrition Research Center
Locations (1):
- USDA, ARS, Western Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mo Z, Huang S, Burnett DJ, Rutledge JC, Hwang DH. Endotoxin May Not Be the Major Cause of Postprandial Inflammation in Adults Who Consume a Single High-Fat or Moderately High-Fat Meal. J Nutr. 2020 May 1;150(5):1303-1312. doi: 10.1093/jn/nxaa003. PMID 32040591